CLINICAL TRIAL: NCT02503267
Title: "Incidence and Consequences of Disorders of Glycosylation in Patients With Conotruncal and Septal Heart Defects" (CARDIoG)
Brief Title: "Incidence and Consequences of Disorders of Glycosylation in Patients With Conotruncal and Septal Heart Defects"
Acronym: (CARDIoG)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Universidad de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIoG
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Congenital Heart Diseases; Conotruncal Defects; Congenital Disorder of Glycosylation; Antithrombin III Deficiency
Keywords: antithrombin III deficiency; congenital heart diseases
MeSH Terms: conditions — Heart Defects, Congenital; Congenital Disorders of Glycosylation; Antithrombin III Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Through the blood sample we will:
  * Identify Antitrombin III deficiency
  * Evaluate the glycosylation degree of different glycoproteins
  * Do a genetic analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with congenital heart disease: patients with congenital heart disease
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention

SUMMARY:
The objective of the study is to investigate congenital disorders of glycosylation in congenital heart diseases without a clear molecular or genetic basis.

DETAILED DESCRIPTION:
Congenital disorders of glycosylation (CDG) are a family of inherited disorders caused by defects in the synthesis of glycans, glycoproteins or other glycoconjugates. Congenital disorders of glycosylation (CDG) are a family of inherited disorders caused by defects in the synthesis of glycans, glycoproteins or other glycoconjugates. Glycosylation of proteins is crucial for a proper organ morphogenesis and for an appropriate coagulation system functioning. The neurological system is commonly affected in this type of disorders but cases of CDG with normal neurological development have been recently described. The group of Experimental Hematology and Clinic Oncology of the University of Murcia (Spain) recently described a rare disorder of glycosylation (ALG12-CDG) as the cause of antithrombin deficiency in a patient of 19 years with a history of repaired ventricular septal defect.

On the other hand, population studies have shown an increased incidence of thromboembolic events in patients with congenital heart disease when compared to the general population. The identified genetic defects involved in the development of congenital heart diseases have variable or incomplete penetrance and in most cases the molecular basis is completely unknown.

The investigators postulate that a CDG might be behind the development of some forms of congenital heart disease and contribute to the greater prevalence of thromboembolic events in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a congenital heart disease with most probability to present a congenital disorder of glycosylation of proteins

Exclusion Criteria:

* Denial of informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250-300 adult patients who are most likely to have a congenital disorder of glycosylation of proteins, such as ventricular and atrial septal defects and especially conotruncal defects
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Disorders of glycosylation | 1 year

SECONDARY OUTCOMES:
Incidence of antithrombin deficiency | 1 year

OTHER OUTCOMES:
Genetical alteractions of disorders of glycosylation | 1 year
Association between disorders of glycosylation and thromboembolic events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron Hospital, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Footitt EJ, Karimova A, Burch M, Yayeh T, Dupre T, Vuillaumier-Barrot S, Chantret I, Moore SE, Seta N, Grunewald S. Cardiomyopathy in the congenital disorders of glycosylation (CDG): a case of late presentation and literature review. J Inherit Metab Dis. 2009 Dec;32 Suppl 1:S313-9. doi: 10.1007/s10545-009-1262-1. Epub 2009 Sep 7. PMID 19757145
- [Background] Gehrmann J, Sohlbach K, Linnebank M, Bohles HJ, Buderus S, Kehl HG, Vogt J, Harms E, Marquardt T. Cardiomyopathy in congenital disorders of glycosylation. Cardiol Young. 2003 Aug;13(4):345-51. PMID 14694955
- [Background] Romano S, Bajolle F, Valayannopoulos V, Lyonnet S, Colomb V, de Barace C, Vouhe P, Pouard P, Vuillaumier-Barrot S, Dupre T, de Keyzer Y, Sidi D, Seta N, Bonnet D, de Lonlay P. Conotruncal heart defects in three patients with congenital disorder of glycosylation type Ia (CDG Ia). J Med Genet. 2009 Apr;46(4):287-8. doi: 10.1136/jmg.2008.057620. No abstract available. PMID 19357119
- [Background] Mitra N, Sinha S, Ramya TN, Surolia A. N-linked oligosaccharides as outfitters for glycoprotein folding, form and function. Trends Biochem Sci. 2006 Mar;31(3):156-63. doi: 10.1016/j.tibs.2006.01.003. Epub 2006 Feb 10. PMID 16473013
- [Background] Lin YS, Liu PH, Wu LS, Chen YM, Chang CJ, Chu PH. Major adverse cardiovascular events in adult congenital heart disease: a population-based follow-up study from Taiwan. BMC Cardiovasc Disord. 2014 Mar 21;14:38. doi: 10.1186/1471-2261-14-38. PMID 24655794
- [Background] de la Morena-Barrio ME, Hernandez-Caselles T, Corral J, Garcia-Lopez R, Martinez-Martinez I, Perez-Duenas B, Altisent C, Sevivas T, Kristensen SR, Guillen-Navarro E, Minano A, Vicente V, Jaeken J, Lozano ML. GPI-anchor and GPI-anchored protein expression in PMM2-CDG patients. Orphanet J Rare Dis. 2013 Oct 20;8:170. doi: 10.1186/1750-1172-8-170. PMID 24139637
- [Background] Martinez-Martinez I, Ordonez A, Navarro-Fernandez J, Perez-Lara A, Gutierrez-Gallego R, Giraldo R, Martinez C, Llop E, Vicente V, Corral J. Antithrombin Murcia (K241E) causing antithrombin deficiency: a possible role for altered glycosylation. Haematologica. 2010 Aug;95(8):1358-65. doi: 10.3324/haematol.2009.015487. Epub 2010 Apr 30. PMID 20435622
- [Background] Aguila S, Martinez-Martinez I, Dichiara G, Gutierrez-Gallego R, Navarro-Fernandez J, Vicente V, Corral J. Increased N-glycosylation efficiency by generation of an aromatic sequon on N135 of antithrombin. PLoS One. 2014 Dec 8;9(12):e114454. doi: 10.1371/journal.pone.0114454. eCollection 2014. PMID 25485983
- [Background] Dorn C, Grunert M, Sperling SR. Application of high-throughput sequencing for studying genomic variations in congenital heart disease. Brief Funct Genomics. 2014 Jan;13(1):51-65. doi: 10.1093/bfgp/elt040. Epub 2013 Oct 3. PMID 24095982